CLINICAL TRIAL: NCT05128253
Title: Characterization of the Platelet Inflammatory Response in NAFL and NASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stefania Basili (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor-Investigator, Stefania Basili, Prof. Stefania Basili, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: 6216
Record Dates: First submitted 2021-07-06; First posted 2021-11-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAFLD
Keywords: platelets; inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous Blood will be centrifuged within 2 hours and plasma and serum samples will be stored at -80°C for further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NASH GROUP: Recruited (n=22) patients with non-alcoholic steatohepatitis.
  Interventions: Other: High fat meal in a subset of patients with NAFL or NASH
- NAFL GROUP: Recruited (n=22) patients with non-alcoholic fatty liver.
  Interventions: Other: High fat meal in a subset of patients with NAFL or NASH

INTERVENTIONS:
Other: High fat meal in a subset of patients with NAFL or NASH — In a subset of NAFL (n=11) and NASH (n=11) patients venous blood samples will also be taken 2 (T0+2h), 4 (T0+4h) and 6 (T0+6h) hours after consumption of a high fat meal.

SUMMARY:
The primary objective of the study is to identify which features of platelet activation promote the inflammatory response that underlies the progression from NAFL to NASH.

Therefore, the investigators plan:

1. To characterize and compare the platelet inflammatory phenotype in NAFL vs NASH patients
2. To study if and how the signaling pathways controlled by ITAM/ITIM-coupled receptors is dysregulated in NAFL vs NASH As a secondary objective the investigators will analyze platelet activation and inflammatory response in a subset of NAFL and NASH patients after 2, 4 and 6 hours from consumption of a high fat meal to test if and how the platelet inflammatory phenotype is promoted by post-prandial plasma lipids.

DETAILED DESCRIPTION:
Background NonAlcoholic Fatty Liver Disease (NAFLD) is one of the most commonly encountered liver disorders worldwide. NAFLD is a spectrum of liver disease including (i) simple hepatic steatosis also called Non-Alcoholic Fatty Liver (NAFL) and (ii) Non-alcoholic SteatoHepatitis (NASH).

When more than 5% hepatic steatosis is present, patients are considered to have NAFL. If steatosis is present along with hepatocyte ballooning degeneration and lobular inflammation, patients are considered to have NASH. About 20% of patients with NAFLD have NASH.

Over time, NAFLD may progress to cirrhosis and ultimately to hepatocellular carcinoma (HCC) with a greater proportion of NASH patients (20%).

Platelets are specialized blood cells that continuously monitor and preserve the integrity of the cardiovascular system. Beyond their well-established role in hemostasis, platelets have been recently shown to actively participate in the inflammatory response and in tissue remodeling, by releasing bioactive molecules and by interacting with leukocytes.

The liver-platelet relationship is very complex. In physiological conditions the liver regulates platelet number by producing thrombopoietin and platelet lifespan by clearing aged platelets. In pathological conditions, increasing evidence demonstrate that platelets have an important role in regulating liver inflammation and chronic disease. Platelet-derived cytokines, such as TGF-β, platelet-derived growth factor-β (PDGF-β), and CXCL4, promote hepatic fibrosis, and platelet count has been used for many years as a surrogate marker of liver fibrosis (FIB-4 index). Recent studies demonstrate that platelet number and platelet aggregation are increased in liver sinusoids of NASH patients. Mechanistic insights provided by mouse models suggest that the role of platelets in NAFLD progression is mediated through the interaction with immune cells. Platelet colonization of the liver is mediated through the interaction with specialized macrophages lining the liver sinusoids (Kupffer cells) and it is a critical step for the recruitment of CD8+ T cells and NKT cells, which drive NASH progression through the release of cytokines and the metabolic reprogramming of hepatocytes. The importance of platelets in the development of NASH and subsequent progression to cirrhosis and HCC has been confirmed in humans by inhibiting platelets with a combination of aspirin and clopidogrel in a small pilot case study.

There is mounting evidence suggesting that distinct signaling pathways regulate the hemostatic and the inflammatory function of platelets. For instance, the platelet ITAM- (GPVI, CLEC2) and ITIM- (PECAM-1, TLT-1) coupled receptors regulate the platelet inflammatory response but have a minor role in hemostasis. Thus, one could envisage targeting the platelet inflammatory response as a strategy to limit the progression of NAFLD, without undermining hemostasis.

Hypotheses The overarching hypothesis of the proposed project is that platelets amplify the inflammatory state that drives the progression from NAFL to NASH.

Platelets participate in the inflammatory response by releasing bioactive compounds and establishing heterotypic interactions with leukocytes. However, these mechanisms in the context of chronic liver disease are poorly understood and have been studied mainly in mice.

Our working model is that platelets docked in the liver of NAFLD patients amplify the inflammatory state by releasing pro-inflammatory cytokines, which in turn recruit and activate leukocytes in the liver sinusoids. Combined stimuli from leukocytes and platelets would then lead to metabolic reprogramming of hepatocytes and progression to NASH. In this context the investigators expect to identify an important role of GPVI and CLEC-2 and their inhibitory counterparts PECAM-1 and TLT-1, which are critically implicated in the regulation of platelet activation at sites of inflammation.

The investigators anticipate that features of the platelet inflammatory response could be both sensitive and sex-specific biomarkers for NASH progression and novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Written informed consent
* Both sexes
* Patients with NAFL and NASH according to EASL Guidelines 2016.

Exclusion Criteria:

* Patients on anti-platelet or anti-coagulant medications
* Reported severe immunosuppression
* Uncontrolled diabetes mellitus type 2 (HbA1c >7.0 %)
* Patients receiving PPAR-gamma and PPAR-alpha agonists
* Uncompensated cirrhosis defined as the presence of at least one of the following features: current or past cirrhosis complications (e.g. ascites, variceal gastrointestinal bleeding, hepatic encephalopathy), the presence of hyperbilirubinaemia (>2 mg/dl), hypoalbuminaemia (<3.2 g/dl), prolonged INR (>1.7), low platelet count, gastroesophageal varices at endoscopy.
* preexisting medical condition with a life expectancy of less than 3 months

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 44 patients (22 with NAFL and 22 NASH) will be enrolled at the Policlinico Umberto I-Sapienza University of Rome, defined according to the EASL Guidelines 2016.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-09-06 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of platelet-leukocyte aggregates (evaluated as median fluorescence intensity -MFI- of platelets bound to leukocytes) in whole blood in patients with NAFLD and NASH | 1 year
  Platelet leukocyte aggregates are a sensitive surrogate marker of platelet activation. The level of platelet-leukocyte aggregates will be measured directly in anticoagulated whole blood, within 30 minutes from withdrawal. By multicolor flow cytometry the investigators will detect the percentage of leukocyte that stain positive for CD41a, a specific marker platelets. The investigators expect to detect a relevant difference in platelet-leukocytes aggregates of 10% between NASH and NAFLD patients.

CONTACTS AND LOCATIONS:
Overall Officials: STEFANIA BASILI, MD, Principal Investigator — SAPIENZA UNIVERSITY- Department of Translational and Precision Medicine
Locations (2):
- Italy (2):
  - Policlinico Umberto Primo - Sapienza University of Rome, Rome
  - Sapienza University of Rome - Policlinico Umberto I Roma, Rome

IPD SHARING:
Plan to Share IPD: No